CLINICAL TRIAL: NCT06874751
Title: Semaglutide Effects on Cardiovascular Outcomes in People With Overweight or Obesity in the Real World
Acronym: SCORE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-8515; U1111-1318-9978 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Overweight; Obesity; Atherosclerotic Cardiovascular Disease (ASCVD)
MeSH Terms: conditions — Overweight; Obesity; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort: Semaglutide Users: Participants age above or equal to (≥) 45 years with overweight or obesity and established ASCVD who initiated semaglutide 2.4 mg (semaglutide 2.4 mg users).
  Interventions: Other: No treatment given
- Cohort: Semaglutide Non-users: Participants age above or equal to (≥) 45 years with overweight or obesity and established ASCVD who are semaglutide 2.4 mg non-users.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given
  Groups: Cohort: Semaglutide Users
Other: No treatment given — No treatment given
  Groups: Cohort: Semaglutide Non-users

SUMMARY:
This is a retrospective database study which includes administrative medical and pharmacy claims linked with clinical and laboratory measurements for patients in the US, to evaluate the effectiveness of once-weekly semaglutide 2.4 mg in reducing the risk of CV and other obesity-related clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with overweight or obesity defined as at least one overweight/obesity indication of a specified body mass index (BMI) above or equal to (≥) 27.0 kilogram per meter square (kg/m^2) and undefined obesity/overweight indications, defined by diagnoses and laboratory values
2. Participants with established ASCVD defined as a diagnosis of MI, diagnosis of ischemic stroke, and/or evidence of peripheral arterial disease
3. Participants who are above or equal to (≥) 45 years old by the end of data availability
4. Participants who initiated semaglutide 2.4 mg on or after the eligibility date and June4, 2021 (semaglutide 2.4 mg users) or participants with no evidence of semaglutide 2.4 mg usage (non-users) during January 1, 2016 to December 31, 2023
5. Participant with continuous insurance enrolment eligibility above or equal to (≥)12 months prior to the index date
6. Participants with re-confirmed overweight/obesity indication during the baseline period

Exclusion criteria:

1. Participants with a diagnosis of chronic or acute pancreatitis
2. Participants with a diagnosis of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
3. Participants with end-stage kidney disease (ESKD) including chronic or intermittent hemodialysis or peritoneal dialysis, kidney transplant, and/or record of estimate glomerular filtration rate less than (<) 15 milliliter per minute per 1.73*meter square (mL/min/1.73m^2)
4. Pregnancy in female participants
5. Participants with evidence of diabetes including more or equal to (≥)2 diagnoses of type 1 diabetes or more or equal to ( ≥) 2 diagnoses of type 2 diabetes on distinct dates, use of a glucose-lowering agent, and/or glycated hemoglobin (HbA1c) laboratory result above or equal to 6.5 percent (%)
6. Use of a glucagon-like peptide-1 (GLP-1) or GLP-1/gastric inhibitory polypeptide (GIP) receptor ago-nist approved for weight management (excluding semaglutide 2.4 mg)
7. Participants with evidence of bariatric surgery

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult participants, age above or equal to 45 years with overweight or obesity and established ASCVD will be included in the study. The eligibility date will be defined as the latest of the following dates: first overweight/ obesity ascertainment, first ASCVD diagnosis, and date participant reached age 45. Then, these participants will be divided into those who initiated semaglutide 2.4 mg (semaglutide 2.4 mg users) and those who did not (non-users).
Sampling Method: Non-Probability Sample
Enrollment: 45456 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Revised 5-Point Major Adverse Cardiovascular Events (MACE-5) (time-to-event) | Index date, earliest of revised MACE-5 and end of follow-up, up to 30 months
  Measured as months
  Occurrence of any of the following individual component events:
  1. Myocardial Infarction (MI)
  2. Stroke
  3. Hospitalization for Heart Failure (HF)
  4. Coronary revascularization
  5. All-cause mortality The event date will be the earliest occurrence of one of the individual components.
Revised 3-Point Major Adverse Cardiovascular Events (MACE-3) (time-to-event) | Index date, earliest of revised MACE-3 and end of follow-up, up to 30 months
  Measured as months
  Occurrence of any of the following individual component events:
  1. MI
  2. Stroke
  3. All-cause mortality The event date will be the earliest occurrence of one of the individual components.

SECONDARY OUTCOMES:
MI (time-to-event) | Index date, earliest of MI and end of follow-up, up to 30 months
  Measured as months
  Participants who were diagnosed of MI (identified using International Classification of Disease, 10th Edition, Clinical Modification [ICD-10-CM] diagnosis codes) observed during an inpatient (IP) visit. The event date will be admission date of the IP visit.
Stroke (time-to-event) | Index date, earliest of stroke and end of follow-up, up to 30 months
  Measured as months
  Participants who were diagnosed of stroke, including both ischemic and hemorrhagic, (identified using ICD-10- CM diagnosis codes) which was observed during an IP visit. The event date will be the admission date of the IP visit.
Hospitalization for HF (time-to-event) | Index date, earliest of hospitalization for HF and end of follow up, up to 30 months
  Measured as months
  Participants who were diagnosed of HF (identified using ICD-10-CM diagnosis codes) observed during an IP visit. The event date will be the first observed admission date of the IP visit.
Coronary revascularization (time-to-event) | Index date, earliest of hospitalization for Coronary revascularization and end of follow up, up to 30 months
  Measured as months
  Participants with evidence of coronary revascularization in any claim (identified using ICD-10-PCS, Current Procedural Terminology [CPT], or Healthcare Common Procedure Coding System [HCPCS] procedure codes). The event date will be the first observed date of coronary revascularization.
All-cause mortality (time-to-event) | Index date, end of follow up, up to 30 months
  Measured as months
  Participants with evidence of death as recorded at the month and year level in KRD and defined as a death record observed within the last month of follow-up. The event date will be the earliest of the end of follow-up (e.g., bariatric surgery within the month of death and last month of follow-up) or the last day of the recorded month of death.
MACE-5 | Index date, earliest of MACE-5 and end of follow-up, up to 30 months
  Measured as months
  Occurrence of any of the following individual component events:
  1. MI
  2. Stroke
  3. Hospitalization for HF
  4. Coronary revascularization
  5. CV-related mortality The event date will be the earliest occurrence of one of the individual components.
MACE-3 | Index date, earliest of MACE-3 and end of follow-up, up to 30 months
  Measured as months
  Occurrence of any of the following individual component events:
  1. MI
  2. Stroke
  3. CV-related mortality The event date will be the earliest occurrence of one of the individual components.
CV-related mortality (time-to-event) | Index date, earliest of MACE-3 and end of follow-up, up to 30 months
  Measured as months
  Partcipants with any claim within ≤30 days before the date of death (i.e., the last day of the recorded month of death, where death is observed in the last month of follow-up) of the following operational definition to indicate a CV-related mortality (identified using ICD-10-CM diagnosis codes): (1) A primary diagnosis of MI (2) A primary diagnosis of ischemic or hemorrhagic stroke (3) A primary diagnosis of HF (4) Evidence of peripheral arterial revascularization, coronary revascularization, CABG, PCI, or carotid intervention in any claim (identified using ICD-10-PCS, CPT, or HCPCS procedure codes).
  (5) A primary diagnosis of CV hemorrhage (excluding hemorrhagic stroke) (6) A primary diagnosis of other CV conditions including unstable angina, sudden cardiac arrest, cardiogenic shock, and other cerebrovascular and CV events.
  The event date will be the earliest of the end of follow-up (e.g., bariatric surgery within the month of death) or the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: https://novonordisk-trials.com

REFERENCES:
- [Derived] Smolderen KG, Mena-Hurtado C, Zhao Z, Michalak W, Faurby M, Smolarz BG, Kosiborod MN, Song J, Chen Y, Boland J, Nanna MG. Lower risk of cardiovascular events in patients initiated on semaglutide 2.4 mg in the real-world: Results from the SCORE study (Semaglutide Effects on Cardiovascular Outcomes in People with Overweight or Obesity in the Real World). Diabetes Obes Metab. 2025 Nov;27(11):6691-6704. doi: 10.1111/dom.70080. Epub 2025 Sep 9. PMID 40926360